CLINICAL TRIAL: NCT07086924
Title: Genetic Variation in TRAF3IP2 (rs13190932) and Its Association With Psoriasis, Psoriatic Arthritis, and Treatment Outcome With Methotrexate
Brief Title: Genetic Variation in TRAF3IP2 (rs13190932)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Fawzia Mohamed Abdelzaher Mohamed, Resident of Dermatology, Venereology and Andrology,Faculty of Medicine, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Genetic variation in TRAF3IP2
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis; Psoriatic Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — Methotrexate; Genetic Variation; Coat Protein Complex I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): About 30 patients suffering from psoriasis
  Interventions: Drug: Methotrexate
- Group B (Active Comparator): About 10 patients suffering from psoriatic arthritis
  Interventions: Drug: Methotrexate
- Group C (Experimental): About 10 healthy control group
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Assessing the response of psoriasis and psoriatic arthritis to Methotrexate. and also Assessing the pharmacogenetic association between TRAF3IP2 ( rs13190932 ) gene Polymorphism in psoriatic and psoriatic arthritis patients taking Methotrexate.
  Other Names: Genetic variation in TRAF3IP2

SUMMARY:
Psoriasis is an immune-mediated inflammatory disease that is highly prevalent worldwide, affecting approximately 2-3% of the world population.

It is characterized by red, scaly plaques that can appear on various parts of the body, causing significant physical and psychological burden to affected individuals.

The Pathogenesis of PsA involves a complex interplay of genetic, immunological, and environmental factors.Genetic studies have identified several susceptibility loci, including HLA-Cw6 and IL23R, which are shared with psoriasis. Additionally, the presence of certain alleles, such as HLA-B27, is associated with a more severe disease course and a higher likelihood of axial involvement.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a chronic systemic inflammatory arthritis that involves both peripheral joints and axial skeleton associated with psoriasis. The extra-articular manifestations and comorbidities are also very common. PsA develops in up to 30% of patients with psoriasis, accounting for an estimated 0.3-1.0% of the general population.

The exact aetiopathogenesis of psoriasis is not completely explained. Pathological mechanism involves skin inflammation and hyperproliferation of keratinocytes induced innate and adaptive immune cells. Genetic, immunological and environmental factors are considered the most important aetiologies . Anti-psoriatic topical preparations, such as those containingcorticosteroids or vitamin D3 analogs (usually calcipotriol [Cal]), are the mainstay of treatment of mild-to-moderate plaque psoriasis. Phototherapy and systemic drugs (administered orally or by injection or infusion) are reserved for more severe or refractory psoriasis.

Methotrexate (MTX) has remained the backbone of the treatment for moderate to severe psoriasis ever since its first use nearly half a century ago. Over the years, its high efficacy, low cost, relative ease of administration and usefulness in concomitant psoriatic arthritis have contributed in making MTX the drug of choice in managing severe psoriasis. Although the majority of patients achieve remission of disease activity with MTX, a significant proportion may experience mild and transient adverse effects. From time to time, various guidelines on the use of MTX have correctly and adequately stressed the need for strict monitoring of haematological and hepatic adverse events.

Characterizing psoriatic arthritis (PsA), mainly as an immune-mediated disease that is also affected by barrier proteins. One new PsA and psoriasis-susceptibility gene, TRAF3IP2, codes for the adaptor protein ACT1 (nuclear factor-κB activator 1), a regulator of the NF-κB pathway involved in IL-17 signaling. We were able to identify the common coding variant p.Asp10Aspn as the disease-causing allele with evidence from association findings at single nucleotide polymorphism (SNP) and haplotype levels, as well as binding studies of ACT1 with its interaction partner TRAF6.

TRAF3 is one of the most versatile members of the TRAF family. It is an intracellular protein that primarily acts as an adaptor protein with a large variety of binding partners. TRAF3 interacting protein 2 (TRAF3IP2), also called CIKS or Act1, is a key intermediate in the normal inflammatory response and is involved in the pathogenesis of various autoimmune and inflammatory diseases .Furthermore, TRAF3IP2 is a protein acting downstream of the IL-17 receptor that binds to and stabilizes mRNAs encoding key inflammatory proteins.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 -70years .
* the severity of cutaneous affection is categorized according to PASI score into PASI 7-12 (moderate severity), and PASI > 12 (severe severity). (15)Confirmed diagnosis: Psoriasis vulgaris (PsV) or psoriatic arthritis (PsA) diagnosed by the Dermatologist or the Rheumatologist.
* Willingness to participate: Signed informed consent.
* Initiating methotrexate (MTX) therapy: For prospective cohort.
* Availability for follow-up: Patients must be willing and able to attend scheduled visit.

Exclusion Criteria:

* Patients with other autoimmune conditions (e.g., rheumatoid arthritis, systemic lupus erythematosus).
* Pregnancy and lactation.
* Patients currently undergoing immunosuppressive or systemic therapies.
* Patients with known genetic disorders affect immune system function.
* Patients with liver or kidney impairment.
* Patients with allergy or contraindication to methotrexate.
* Patients with active or uncontrolled infections, including chronic infections like tuberculosis.
* Previous genetic analysis Patients who have previously undergone genetic analysis for the TRAF3IP2 gene polymorphism (rs13190932).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Treatment of Psoriasis and Psoriatic arthritis | 3 months
  Treatment the patients whom suffering from Psoriasis and Psoriatic arthritis and Assessment of clinical improvement to methotrexate therapy according to: PASI score into PASI 50: means 50% reduction in PASI score - an acceptable measure of efficacy for secondary endpoints in psoriasis clinical trials PASI 75: means 75% reduction in PASI score - standard efficacy measure used in most psoriasis clinical studies1 PASI 90: means 90% reduction in PASI score (almost clear skin) PASI 100: means Completely clear skin.
Evalaute the effect of treatment with Methotrexate | 3 months
  Evaluate the effect of treatment with methotrexate therapy (15 mg per week) on the level of serum TRAF3IP2( rs13190932 ) gene Polymorphism on the Participants whom suffering from Psoriasis and Psoriatic arthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Eisa Mohammed Hegazy, Professor, Study Chair — Dermatology,Venereology,and Andrology Department,Faculty of Medicine,South Valley University, Egypt
Locations (1):
- Qena Hospital, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided